CLINICAL TRIAL: NCT04713865
Title: The Acute and Long-term Clinical Outcome of Self- Expandable Stent in Complex Proximal Superficial Femoral Artery Lesions Involving the Femoral Bifurcation
Status: Not yet recruiting | Type: Observational
Sponsor: Qingdao Hiser Medical Group (Other)
Responsible Party: Sponsor
Other Study IDs: the Sent-FP study
Record Dates: First submitted 2021-01-15; First posted 2021-01-19 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-01

CONDITIONS: Common Femoral Artery Occlusive Disease
Keywords: Common femoral artery occlusive disease; The bare metal stent; profound femoral artery patency

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- PFA slightly jailed by proximal SFA stent(100 pts)
  Interventions: Procedure: endovascular treatment
- PFA moderately jailed by proximal SFA stent(100 pts)
  Interventions: Procedure: endovascular treatment
- PFA totally jailed by proximal SFA stent (100pts)
  Interventions: Procedure: endovascular treatment

INTERVENTIONS:
Procedure: endovascular treatment — The bare metal stent covers the deep femoral artery lower than 50%
  Groups: PFA slightly jailed by proximal SFA stent(100 pts)
Procedure: endovascular treatment — The bare metal stent covers the deep femoral artery in 50-90%
  Groups: PFA moderately jailed by proximal SFA stent(100 pts)
Procedure: endovascular treatment — The bare metal stent totally covers the deep femoral artery
  Groups: PFA totally jailed by proximal SFA stent (100pts)

SUMMARY:
The stent-FP study investigates the impact of coverage of profound femoral artery (PFA) by bare metal stent deployed in proximal superficial femoral artery (SFA) lesions. 300 patients with femoral bifurcation lesions will be included and divided into 3 groups according to the location of proximal stent edge. The primary endpoint of the study is major adverse events and freedom from target lesion revascularization at 48 months. Secondary endpoints include primary patency of PFA and bare metal stent at 1,6, 12,24,36and 48 month, MAE and F -TLR at 1,6, 12,24,36 month.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with chronic atherosclerosis obliterans aged over 18 years
2. Patients presenting Rutherford classification from 2-5
3. Patients is willing to follow-up on time
4. Patient has a life expectancy of at least 24 months
5. Prior to enrolment, the guidewire has crossed target lesion
6. De novo lesions located in the femoral artery bifurcation (5mm between distal CFA and proximal SFA), need for primary bare metal stent implantation
7. There is a patent deep femoral artery demonstrated by angiography
8. If the first-time endovascular treatment is failure, patients undergo endovascular treatment successfully at the second time, the patients can still be enrolled （9）For patients with aortoiliac artery lesions, they can be enrolled after the successful reconstruction of aortoiliac artery .

(10) The lower extremity artery needs to have a healthy runoff of no less than 10 cm above the ankle, and at least one healthy dorsalis pedis artery, medial or lateral plantar artery connected with the digital artery below the ankle (11) Informed consent signed by patients

Exclusion Criteria:

1. Patients who are known to be allergic to heparin, low molecular weight heparin, contrast agents, etc.
2. In the past 3 months, they have participated in other drugs that interfere with this clinical trial or patients in clinical trials of medical devices
3. Pregnant and lactating women
4. Patients with other diseases that may make the trial difficult or significantly shorten the patient's life expectancy (<2 years), such as tumors, severe liver disease, cardiac insufficiency, etc or patients whose life expectancy is less than 24 months (24 months of follow-up are required)
5. Patients with acute arterial thrombosis or embolism at the target lesion site.
6. Patients who underwent stent implantation in common femoral artery previously

(8) Use of thrombectomy, atherectomy or laser devices during procedure (9) Previous open surgery in the same limb . (10) Patients with deep femoral artery totally occlusion

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patiens with De novo lesions located in the femoral artery bifurcation (5mm between distal CFA and proximal SFA), need for primary bare metal stent implantation
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-08-18 (Estimated); Primary Completion 2023-08-17 (Estimated); Study Completion 2026-08-17 (Estimated)

PRIMARY OUTCOMES:
Major adverse events and freedom from target lesion revascularization | post-interventional 48 months
  Major adverse events and freedom from target lesion revascularization at 48 months

SECONDARY OUTCOMES:
primary patency of PFA and bare metal stent | post-interventional 1,6, 12,24,36 and 48 month
  primary patency of PFA and bare metal stent at 1,6, 12,24,36 and 48 month
MAE | post-interventional 1,6, 12,24,36 month
  Major adverse events at 1,6, 12,24,36 month
F -TLR | post-interventional 1,6, 12,24,36 month
  freedom from target lesion revascularization at 1,6, 12,24,36 month